CLINICAL TRIAL: NCT06955468
Title: Development of a Bidirectional Priming Intervention for Goals-of-care Communication in Oncology
Brief Title: Evaluating a Bidirectional Priming Intervention for Goals-of-care Communication in Oncology
Acronym: Prime GOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 26924
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancers; Gastrointestinal Cancers
Keywords: Communication
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will complete a survey prior to hospital discharge. Their responses will be shared with each participant's outpatient oncology team.
  Interventions: Behavioral: Priming Survey
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Priming Survey — 13-item priming survey assessing patients' goals, treatment preferences, and disease understanding.
  Arms: Intervention

SUMMARY:
This pilot study will evaluate whether an intervention aimed at hospitalized patients with advanced lung and gastrointestinal cancers can help facilitate goals-of-care (GOC) communication with their oncologists after discharge.

While GOC communication is a recommended component of routine oncology care, many patients with solid cancers do not have the opportunity to talk with their oncologist about their goals and end-of-life preferences. Prior research has shown that a systematic method of prompting GOC communication with at-risk patients would address a key barrier to timely GOC communication and ensure that patients receive care that is in line with their personal preferences.

This trial will enroll 80 participants, who will be randomized 1:1 to either an intervention or a control group. Participants in the intervention group will complete a short survey regarding their goals, preferences, and disease understanding. Survey responses will be shared with each participant's outpatient oncology team. Oncologists will subsequently receive a nudge in the electronic medical record reminding them of key survey responses and encouraging them to discuss them at the patient's first clinic visit after hospital discharge.

The primary feasibility outcome is intervention completion rate and the primary clinical outcome is GOC documentation within 30 days of discharge in the intervention group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Unplanned admission to the HUP Solid Oncology service;
2. Underlying diagnosis of advanced lung or GI cancer, defined as metastatic or locally advanced disease;
3. Anticipated discharge within the next 72h; and
4. Primary oncologist is based at HUP; or
5. Family member/caregiver of a patient meeting the above 4 criteria.

Exclusion Criteria:

1. Unable to complete survey in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Intervention Completion Rate | From enrollment to 30 days after hospital discharge
  The primary feasibility outcome is intervention completion rate, defined as successful completion of the survey, response sharing, and electronic medical record nudge for all participants assigned to the intervention arm.
GOC Documentation | From enrollment to 30 days after hospital discharge
  The presence of outpatient goals-of-care documentation in the electronic medical record within 30 days of hospital discharge as determined by manual review.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No